CLINICAL TRIAL: NCT06620237
Title: Pivotal Study of the Amvia Pacemaker and Solia CSP S Pacing Lead on Conduction System Pacing
Brief Title: BIO|MASTER.CSP Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BA113
Record Dates: First submitted 2023-02-08; First posted 2024-10-01 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Pacing, Artificial; Cardiac Pacemaker, Artificial; Cardiac Resynchronization Therapy Devices; Bradycardia; Conduction Disorder; Conduction Defect, Cardiac; Heart Failure
Keywords: Conduction system pacing (CSP); Left bundle branch area pacing (LBBAP)
MeSH Terms: conditions — Bradycardia; Arrhythmias, Cardiac; Cardiac Conduction System Disease; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LBBAP Amvia (No Intervention): All patients with successful implantation of Amvia pacemaker and a lead in a position intended for LBBA pacing.
- LBBAP Solia CSP S (Experimental): All patients with successful implantation of a Solia CSP S lead in LBB area. Additionally, all patients with a non-successful Solia CSP S implantation attempt in which an ADE (adverse device effect) or SADE (serious adverse device effect) related to the Solia CSP S lead occurred.
  Interventions: Device: Implantation of the Solia CSP S pacing lead for LBBAP

INTERVENTIONS:
Device: Implantation of the Solia CSP S pacing lead for LBBAP — Left bundle branch area pacing using a Solia CSP S lead
  Arms: LBBAP Solia CSP S

SUMMARY:
The goal of this clinical study is to test the clinical safety and performance of the Amvia pacemakers and the Solia CSP S lead when used for left bundle branch area pacing (LBBAP). The patient population consist of patients with cardiac pacemaker indication or cardiac resynchronization therapy indication and intended for implantation of a system with left bundle branch area stimulation. Participants will visit sites at enrollment in the study, at implantation and pre-hospital discharge, 1-, 6- and 12-month follow-up visits. Additional annual follow-up(s) may apply until study termination after regulatory approval of Solia CSP S. The total duration of the clinical investigation is expected to be until September 2027, with last patient out (LPO). During the visits the regular pacemaker and lead measurement are performed. A 12-lead ECG is recorded to document intrinsic and ventricularly paced heart rhythm to assess left bundle branch area pacing. Programming of the pacemakers will be done according to the participant´s therapeutical needs.

The study will be conducted in approximately 18 sites in Europe, Australia and New Zealand where more than one physician per site are expected to participate.

ELIGIBILITY:
Inclusion Criteria:

For patient enrollment in the study all of the following inclusion criteria have to be fulfilled at the time of enrollment:

* Standard indication for de novo pacemaker implantation or cardiac resynchronization therapy (CRT)
* Patient is intended for implantation of a pacemaker or CRT-P system with left bundle branch area stimulation
* Ability to understand the nature of the study
* Ability and willingness to perform all follow-up visits at the study site
* Ability and willingness to use the CardioMessenger and acceptance of the BIOTRONIK Home Monitoring concept

Exclusion Criteria:

Enrollment of a patient is not permitted if at least one of the following criteria is fulfilled:

* Planned cardiac surgical procedures or interventional measures other than the study procedure within the next 12 months
* Expected to receive heart transplantation or ventricular assist device within 12 months
* Life-expectancy less than 12 months
* Pregnant or breast feeding
* Age less than 18 years
* Participation in another interventional clinical investigation (according to the definition given in the CIP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Amvia related SADE-d free rate | 6 months (183 days) after implantation
  rate of serious adverse device effects possible, probable or causal related to the Amvia pacemaker
Solia CSP S related SADE-d free rate | 6 months (183 days) after implantation
  rate of serious adverse device effects possible, probable or causal related to the Solia CSP S lead

SECONDARY OUTCOMES:
Amvia related SADE-d free rate | 12 months (365 days) after implantation
  Rate of serious adverse device effects possible, probable or causal related to the Amvia pacemaker
Solia CSP S related SADE-d free rate | 12 months (365 days) after implantation
  Rate of serious adverse device effects possible, probable or causal related to the Solia CSP S lead
Rate of successful acute CSP implantation of Solia CSP S | At the day of implantation
  All implantations, in which the investigator decides to leave the Solia CSP S pacing lead permanently in the conduction system, are counted as acute success.
Sensing performance | At the day of implantation and at the date of each in-office patient follow-up visit (1-, 6-, 12-month follow-up, and annual follow-up*) * please refer to study duration in study description section
  Investigators will be asked whether the sensing is adequate (yes/no decision)
Pacing performance | At the day of implantation and at the date of each in-office patient follow-up visit (1-, 6-, 12-month follow-up, and annual follow-up*) * please refer to study duration in study description section
  Investigators will be asked whether the pacing is adequate (yes/no decision)
Physiologic ventricular excitation | At the day of implantation and at the date of each in-office patient follow-up visit (1-, 6-, 12-month follow-up, and annual follow-up*) * please refer to study duration in study description section
  Investigators are asked to assess whether pacing in the left bundle branch area is still present based on the 12-lead ECG recording
Mid-term change in LVEF | At baseline, at the 6-month follow-up, at the 12-month follow-up and at all following annual in-office follow-ups*, if applicable; * please refer to study duration in study description section
  Collection of left ventricular ejection fraction (LVEF) values
Mid-term change in LVESV | At baseline, at the 6-month follow-up, at the 12-month follow-up and at all following annual in-office follow-ups*, if applicable; * please refer to study duration in study description section
  Collection of left ventricular ejection systolic volume (LVESV) values
Mid-term change in quality of life, EQ-5D-5L (EuroQol) questionnaire | At baseline after patient enrollment prior to implantation, at the date of 6-month follow-up, at the 12-month follow-up and at all following annual in-office follow-ups*, if applicable; * please refer to study duration in study description section
  Collection of health-related quality of life questionnaires from the patient to monitor mid-term changes in the quality of life, analysis and reporting according to EuroQol methodology
Mid-term change in quality of life, SF-36 (Short Form Health Survey) questionnaire | At baseline after patient enrollment prior to implantation, at the date of 6-month follow-up, at the 12-month follow-up and at all following annual in-office follow-ups*, if applicable; * please refer to study duration in study description section
  Collection of health-related quality of life questionnaires from the patient to monitor mid-term changes in the quality of life, analysis and reporting according to item short form health survey (SF-36) standard methodology

CONTACTS AND LOCATIONS:
Overall Officials: Jan De Pooter, MD, PhD, Study Chair — University Hospital Ghent, Gent (Belgium)
Locations (14):
- Australia (3):
  - Integral Healthcare, Adelaide
  - Victorian Heart Hospital, Clayton
  - Lyell McEwin Hospital, Elizabeth Vale
- Belgium (4):
  - AZ Sint-Jan, Bruges
  - Grand Hôpital de Charleroi, Charleroi
  - UZ Gent - Universitair Ziekenhuis Gent, Ghent
  - Clinique Saint-Pierre Ottignies, Ottignies
- France (4):
  - Hopital de la Timone (CHU La Timone), Marseille
  - Centre Hospitalier Metz-Thionville, Metz
  - Hôpital privé du Confluent, Nantes
  - Hôpital Haut Lévêque (CHU), Pessac
- Netherlands (2):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Catharina Ziekenhuis, Eindhoven
- Auckland City Hospital, Grafton, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data may be shared with qualified healthcare practitioners or academic researchers upon request and with permission of BIOTRONIK. Requests shall be sent to the Clinical Research Department of BIOTRONIK.